CLINICAL TRIAL: NCT00358826
Title: Clinical Study Protocol No. VIA-2291-01, A Phase 2 Randomized, Double-blind, Parallel-group, Placebo-controlled, Dose-ranging Study of the Effect of VIA-2291 on Vascular Inflammation in Patients After an Acute Coronary Syndrome Event
Brief Title: Study Effect of VIA-2291 on Vascular Inflammation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tallikut Pharmaceuticals, Inc. (Industry)
Collaborators: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIA-2291-01
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Results first posted 2012-07-23 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — atreleuton

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- VIA-2291 25 mg (Experimental): VIA-2291 25 mg
  Interventions: Drug: VIA-2291
- VIA-2291 50 mg (Experimental): VIA-2291 50 mg
  Interventions: Drug: VIA-2291
- VIA-2291 100 mg (Experimental): VIA-2291 100 mg
  Interventions: Drug: VIA-2291
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIA-2291 — oral dosing, 1 time daily for 12 or 24 weeks
  Other Names: atreleuton
  Arms: VIA-2291 100 mg; VIA-2291 25 mg; VIA-2291 50 mg
Drug: Placebo — oral dosing, 1 time daily for 12 or 24 weeks
  Arms: Placebo

SUMMARY:
This is a dose ranging study to compare the effect of VIA-2291 vs. Placebo on various inflammatory biomarkers in patients with recent acute coronary events

DETAILED DESCRIPTION:
This is a Phase II, randomized, double-blind, placebo-controlled study of the effect of VIA-2291 on atherosclerotic vascular inflammation

ELIGIBILITY:
Inclusion Criteria:

* Female patients are to be of non-childbearing potential
* Patient has suffered an ST elevation myocardial infarction (MI), non-ST elevation MI, or unstable angina 21 days (±3 days) prior to study randomization
* Patient has documented coronary artery disease

Exclusion Criteria:

* Renal insufficiency defined as creatinine >1.5 x upper limit of normal (ULN)
* Cirrhosis, recent hepatitis, ALT >1.5 x ULN or ALT > 1 x ULN and at least one other liver function test
* Uncontrolled diabetes mellitus within 1 month prior to study screening
* Congestive heart failure (CHF) defined by the New York Heart Association as functional Class III or IV
* Previous coronary artery bypass graft (CABG) surgery
* Planned additional cardiac intervention
* Recurrence of ST elevation MI, non-ST elevation MI, or unstable angina less than 18 days prior to randomization
* Current atrial fibrillation, atrial flutter, or frequent premature ventricular contractions
* Acetaminophen use in any form in the 7 days before enrollment

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2006-07; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Taub, MD, Study Director — VIA Pharmaceuticals
Locations (12):
- United States (5):
  - MIMA Century Research Associates, Melbourne, Florida
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Victoria Heart and Vascular Center, Victoria, Texas
- Canada (7):
  - Foothills Medical Center, Calgary, Alberta
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - Queen Elizabeth II HSC, Halifax, Nova Scotia
  - Montreal Heart Institute, Montreal, Quebec
  - Notre Dame Hospital, Montreal, Quebec
  - Hospital Sacre-Coeur, Montreal, Quebec
  - Constituante Centre Hospitalier Regional De Lanaudiere, Saint-Charles-Borromée, Quebec

REFERENCES:
- [Background] Tardif JC, L'allier PL, Ibrahim R, Gregoire JC, Nozza A, Cossette M, Kouz S, Lavoie MA, Paquin J, Brotz TM, Taub R, Pressacco J. Treatment with 5-lipoxygenase inhibitor VIA-2291 (Atreleuton) in patients with recent acute coronary syndrome. Circ Cardiovasc Imaging. 2010 May;3(3):298-307. doi: 10.1161/CIRCIMAGING.110.937169. Epub 2010 Feb 27. PMID 20190281
- [Derived] Matsumoto S, Ibrahim R, Gregoire JC, L'Allier PL, Pressacco J, Tardif JC, Budoff MJ. Effect of treatment with 5-lipoxygenase inhibitor VIA-2291 (atreleuton) on coronary plaque progression: a serial CT angiography study. Clin Cardiol. 2017 Apr;40(4):210-215. doi: 10.1002/clc.22646. Epub 2016 Nov 24. PMID 27883201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients had an Acute Coronary Syndrome (ACS) within 3 weeks prior to randomization
Pre-assignment Details: Subset of patients agreed to participate in a Multi-Detector Computed Tomography (MDCT) substudy for an additional 12 weeks of treatment for a total of 24 weeks
Groups:
- VIA-2291 25 mg: VIA-2291, 25 mg, oral dosing, daily, 12 weeks
- VIA-2291 50 mg: VIA-2291, 50 mg, oral dosing, daily, 12 weeks
- VIA-2291 100 mg: VIA-2291, 100 mg, oral dosing, daily, 12 weeks
- Placebo: Matching Placebo, 12 weeks
- VIA-2291 25 mg MDCT Substudy: VIA-2291, 25 mg, oral dosing, daily, 24 weeks
- VIA-2291 50 mg MDCT Substudy: VIA-2291, 50 mg, oral dosing, daily, 24 weeks
- VIA-2291 100 mg MDCT Substudy: VIA-2291, 100 mg, oral dosing, daily, 24 weeks
- Placebo MDCT Substudy: Matching Placebo, 24 weeks
Period: Core Study
Arm/Group | VIA-2291 25 mg | VIA-2291 50 mg | VIA-2291 100 mg | Placebo | VIA-2291 25 mg MDCT Substudy | VIA-2291 50 mg MDCT Substudy | VIA-2291 100 mg MDCT Substudy | Placebo MDCT Substudy
Started | 49 | 46 | 44 | 52 | 0 | 0 | 0 | 0
Completed | 46 | 41 | 42 | 50 | 0 | 0 | 0 | 0
Not Completed | 3 | 5 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: MDCT Substudy
Arm/Group | VIA-2291 25 mg | VIA-2291 50 mg | VIA-2291 100 mg | Placebo | VIA-2291 25 mg MDCT Substudy | VIA-2291 50 mg MDCT Substudy | VIA-2291 100 mg MDCT Substudy | Placebo MDCT Substudy
Started | 0 | 0 | 0 | 0 | 25 | 22 | 19 | 27
Completed | 0 | 0 | 0 | 0 | 24 | 20 | 19 | 27
Not Completed | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Matching Placebo, oral dosing, 12 weeks
- Total: Total of all reporting groups
Arm/Group | VIA-2291 25 mg | VIA-2291 50 mg | VIA-2291 100 mg | Placebo | Total
Number analyzed (Participants) | 49 | 46 | 44 | 52 | 191
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 38 | 35 | 35 | 41 | 149
  >=65 years | 11 | 11 | 9 | 11 | 42
Age Continuous [Mean (Standard Deviation); unit: years] | 56.4 (9.54) | 57.3 (10.01) | 57.6 (9.44) | 56.6 (9.78) | 57.0 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 6 | 11 | 30
  Male | 41 | 41 | 38 | 41 | 161
Region of Enrollment [Number; unit: participants]
  Canada | 34 | 33 | 31 | 34 | 132
  United States | 15 | 13 | 13 | 18 | 59

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on ex Vivo Leukotriene B4 Synthesis in Whole Blood
Time Frame: Baseline and 12 weeks
Population: Core Study Evaluable Population
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | VIA-2291 25 mg | VIA-2291 50 mg | VIA-2291 100 mg | Placebo
Number analyzed (Participants) | 43 | 36 | 38 | 45
pg/mL | -88126 (29.95) [-100056 to -76196] | -95703 (31.01) [-108810 to -82597] | -122668 (7.01) [-135359 to -109976] | -20843 (174.12) [-32509 to -9179]
Statistical Analysis 1: Comparison: VIA-2291 25 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Adjusted using Dunnett's method; The model included treatment effect, with baseline value as a covariate
Statistical Analysis 2: Comparison: VIA-2291 50 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Adjusted using Dunnett's method; The model included treatment effect, with baseline value as a covariate
Statistical Analysis 3: Comparison: VIA-2291 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Adjusted using Dunnett's method; The model included treatment effect, with baseline value as a covariate

2. Secondary Outcome: Change From Baseline in Leukotriene E4 (LTE4)
Description: Urinary LTE4 is expressed in pg per mg Creatinine (pg/mg Cr) to normalize for renal excretion rate
Time Frame: Baseline and 12 weeks
Population: Core Study Evaluable Population
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mg Cr
Arm/Group | VIA-2291 25 mg | VIA-2291 50 mg | VIA-2291 100 mg | Placebo
Number analyzed (Participants) | 42 | 38 | 35 | 44
pg/mg Cr | -26.8 [-39.3 to -14.4] | -38.6 [-51.7 to -25.5] | -56.5 [-70.2 to -42.9] | 8.4 [-3.8 to 20.6]
Statistical Analysis 1: Comparison: VIA-2291 25 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Adjusted using Dunnett's method; The model included treatment effect, with baseline value as a covariate
Statistical Analysis 2: Comparison: VIA-2291 50 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Adjusted using Dunnett's method; The model included treatment effect, with baseline value as a covariate
Statistical Analysis 3: Comparison: VIA-2291 100 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — Adjusted using Dunnett's method; The model included treatment effect, with baseline value as a covariate

3. Secondary Outcome: Change From Baseline in High Sensitivity C-reactive Protein (hsCRP) - Core Study
Time Frame: Baseline and 12 weeks
Population: Evaluable Population
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | VIA-2291 25 mg | VIA-2291 50 mg | VIA-2291 100 mg | Placebo
Number analyzed (Participants) | 44 | 38 | 38 | 48
mg/L | -0.2 [-1.1 to 0.4] | -0.1 [-1.9 to 0.1] | -0.3 [-0.8 to 0.1] | -0.2 [-0.9 to 0.1]
Statistical Analysis 1: Comparison: VIA-2291 25 mg vs Placebo; Test type: Superiority or Other; p = 0.656, ANCOVA — Adjusted using Dunnett's method
Statistical Analysis 2: Comparison: VIA-2291 50 mg vs Placebo; Test type: Superiority or Other; p = 0.863, ANCOVA — Adjusted using Dunnett's method
Statistical Analysis 3: Comparison: VIA-2291 100 mg vs Placebo; Test type: Superiority or Other; p = 0.996, ANCOVA — Adjusted using Dunnett's method

4. Other Pre Specified Outcome: Change From Baseline in High Sensitivity C-reactive Protein (hsCRP) - MDCT Substudy
Time Frame: Baseline and 24 weeks
Population: Evaluable Population of the MDCT substudy
Measure: Median (Inter-Quartile Range); unit: mg/L
Groups:
- Placebo MDCT Substudy: Matching Placebo, oral dosing, 24 weeks
Arm/Group | VIA-2291 25 mg MDCT Substudy | VIA-2291 50 mg MDCT Substudy | VIA-2291 100 mg MDCT Substudy | Placebo MDCT Substudy
Number analyzed (Participants) | 23 | 20 | 18 | 27
mg/L | -0.4 [-1.2 to 0.3] | -0.2 [-3.7 to 0.2] | -0.4 [-3.9 to -0.2] | 0.0 [-0.5 to 1.2]
Statistical Analysis 1: Comparison: VIA-2291 25 mg MDCT Substudy vs Placebo MDCT Substudy; Test type: Superiority or Other; p = 0.331, ANCOVA — Adjusted using Dunnett's method
Statistical Analysis 2: Comparison: VIA-2291 50 mg MDCT Substudy vs Placebo MDCT Substudy; Test type: Superiority or Other; p = 0.606, ANCOVA — Adjusted using Dunnett's method
Statistical Analysis 3: Comparison: VIA-2291 100 mg MDCT Substudy vs Placebo MDCT Substudy; Test type: Superiority or Other; p < 0.001, ANOVA — Adjusted using Dunnett's method

5. Other Pre Specified Outcome: Change From Baseline in Noncalcified Plaque Volume
Time Frame: Baseline and 24 weeks
Population: Evaluable Population
Measure: Least Squares Mean (95% Confidence Interval); unit: mm^3
Arm/Group | VIA-2291 25 mg MDCT Substudy | VIA-2291 50 mg MDCT Substudy | VIA-2291 100 mg MDCT Substudy | Placebo MDCT Substudy
Number analyzed (Participants) | 7 | 8 | 7 | 12
mm^3 | -1.55 [-5.62 to 2.51] | -5.6 [-9.49 to -1.71] | 0.15 [-3.84 to 4.14] | 2.83 [-0.18 to 5.84]
Statistical Analysis 1: Comparison: VIA-2291 25 mg MDCT Substudy vs Placebo MDCT Substudy; Test type: Superiority or Other; p = 0.22, ANCOVA — Dunnett test compared with Placebo
Statistical Analysis 2: Comparison: VIA-2291 50 mg MDCT Substudy vs Placebo MDCT Substudy; Test type: Superiority or Other; p < 0.005, ANCOVA — Dunnett test compared with Placebo
Statistical Analysis 3: Comparison: VIA-2291 100 mg MDCT Substudy vs Placebo MDCT Substudy; Test type: Superiority or Other; p = 0.60, ANCOVA — Dunnett test compared with Placebo

6. Other Pre Specified Outcome: Change From Baseline in Mean Plaque Density
Description: Plaque density is expressed in Hounsfield Units (HU)
Time Frame: Baseline and 24 weeks
Population: Evaluable Population
Measure: Least Squares Mean (95% Confidence Interval); unit: HU
Arm/Group | VIA-2291 25 mg | VIA-2291 50 mg | VIA-2291 100 mg | Placebo
Number analyzed (Participants) | 7 | 8 | 7 | 12
HU | 19.11 [-1.51 to 39.74] | 7.39 [-11.96 to 26.74] | 12.22 [-8.38 to 32.82] | 12.42 [-3.32 to 28.17]
Statistical Analysis 1: Comparison: VIA-2291 25 mg vs Placebo; Test type: Superiority or Other; p = 0.92, ANCOVA — Dunnett test compared with Placebo
Statistical Analysis 2: Comparison: VIA-2291 50 mg vs Placebo; Test type: Superiority or Other; p = 0.96, ANCOVA — Dunnett test compared with Placebo
Statistical Analysis 3: Comparison: VIA-2291 100 mg vs Placebo; Test type: Superiority or Other; p = 1.00, ANCOVA — Dunnett test compared with Placebo

7. Other Pre Specified Outcome: Change From Baseline in Percent Stenosis
Time Frame: Baseline and 24 weeks
Population: Evaluable Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage
Arm/Group | VIA-2291 25 mg | VIA-2291 50 mg | VIA-2291 100 mg | Placebo
Number analyzed (Participants) | 7 | 8 | 7 | 12
Percentage | -0.11 [-8.24 to 8.03] | 11.45 [3.73 to 19.17] | 2.36 [-5.7 to 10.42] | 1.19 [-4.95 to 7.32]
Statistical Analysis 1: Comparison: VIA-2291 25 mg vs Placebo; Test type: Superiority or Other; p = 0.99, ANCOVA — Dunnett test compared with Placebo
Statistical Analysis 2: Comparison: VIA-2291 50 mg vs Placebo; Test type: Superiority or Other; p = 0.11, ANCOVA — Dunnett test compared with Placebo
Statistical Analysis 3: Comparison: VIA-2291 100 mg vs Placebo; Test type: Superiority or Other; p = 0.99, ANCOVA — Dunnett test compared with Placebo

ADVERSE EVENTS:
Time Frame: 12 weeks for Core Study and 24 weeks for MDCT substudy
Arm/Group | VIA-2291 25 mg | VIA-2291 50 mg | VIA-2291 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 4/49 | 3/46 | 7/44 | 5/52
Other Adverse Events (participants affected / at risk) | 42/49 | 43/46 | 42/44 | 45/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | VIA-2291 25 mg (N=49) | VIA-2291 50 mg (N=46) | VIA-2291 100 mg (N=44) | Placebo (N=52)
Angina Unstable (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0/0 (0) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac Chest Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis Ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accelerated Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal Detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VIA-2291 25 mg (N=49) | VIA-2291 50 mg (N=46) | VIA-2291 100 mg (N=44) | Placebo (N=52)
Fatigue (General disorders) | 4 (4) | 6 (6) | 7 (7) | 5 (5)
Non-cardiac Chest Pain (General disorders) | 5 (5) | 3 (3) | 4 (4) | 4 (4)
Chest pain (General disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4) | 5 (5) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 3 (3) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 5 (5) | 5 (5) | 6 (6)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 7 (7) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 7 (7) | 2 (2)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 4 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 1 (1) | 2 (2)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (4) | 1 (1)
Dspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 4 (4) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 4 (4) | 0 (0)
Angina Pectoris (Cardiac disorders) | 3 (3) | 8 (8) | 7 (7) | 5 (5)
Nasopharyngitis (Infections and infestations) | 1 (1) | 5 (5) | 0 (0) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 5 (5) | 2 (2) | 4 (4) | 7 (7)
Alanine Aminotransferase Increased (Investigations) | 5 (5) | 1 (1) | 1 (1) | 3 (3)
Blood Glucose Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hypertension (Vascular disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 4 (4) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented as a joint, multi-center publication.